CLINICAL TRIAL: NCT00474383
Title: A Phase II Open Label Study of CB7630 (Abiraterone Acetate) in Patients With Advanced Prostate Cancer Who Have Failed Androgen Deprivation and Docetaxel-Based Chemotherapy
Brief Title: An Safety and Efficacy Study of Abiraterone Acetate in Participants With Advanced Prostate Cancer Who Failed Androgen Deprivation and Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016915; COU-AA-003; COU-AA-003EXT; NCT01798615 (Other: ClinicalTrials.gov Identifier); NCT01798615 (obsolete NCT alias)
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; CB7630; Abiraterone acetate; Glucocorticoid; Prednisone; Prednisolone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): Abiraterone acetate 1000 milligram (mg) tablet or capsule will be administered orally, once daily continuously in 28-day cycle up to disease progression, death, or end of study, along with prednisone/prednisolone 5 mg tablet orally twice daily or dexamethasone 0.5 mg tablet orally once daily.
  Interventions: Drug: Abiraterone acetate; Drug: Glucocorticoid

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000 milligram (mg) capsule or tablet will be administered orally, once daily continuously in 28-day cycle up to disease progression, death, or end of study.
Drug: Glucocorticoid — Prednisone/prednisolone 5 mg tablet orally twice daily/dexamethasone 0.5 mg tablet orally once daily continuously in 28-day cycle up to disease progression, death, or end of study.

SUMMARY:
The purpose of this study is to assess the anti-tumor activities and safety of abiraterone acetate in participants with prostate cancer (a disease in which cells in the prostate gland [a gland in the male reproductive system found below the bladder and in front of the rectum] become abnormal and start to grow uncontrollably, forming tumors) who have failed taxane (docetaxel)-based chemotherapy.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single arm, multicenter (when more than one hospital or medical school team work on a medical research study) study to evaluate the anti-tumor activities and safety of abiraterone acetate in participants with cancer who have failed taxane (docetaxel)-based chemotherapy. Abiraterone acetate 1000 milligram (mg) tablet or capsule will be administered orally (by mouth), once daily after an overnight fast until disease progression, lack of disease response after six 28-day cycles of treatment, or when unacceptable toxicity is encountered. Participants will be treated for up to 12 cycles. All participants will receive a concurrent low-dose glucocorticoid (such as prednisone 5 mg tablet twice daily/prednisolone 0.5 mg tablet once daily). Treatment will be continued in responding participants until death, or disease progression, or end of the study (which is Week 148). Efficacy will primarily be assessed through prostate specific antigen response according to Prostate Specific Antigen Working Group (PSAWG) criteria. Participants' safety will be monitored throughout the study. Participants who have completed 12 cycles of abiraterone acetate treatment, and continue to receive clinical benefit from such treatment, will be eligible to enter the extension study. Participants who enter the extension study will continue taking abiraterone acetate at the dose they were receiving at the end of the main study together with low-dose glucocorticoid. Efficacy and safety will be monitored throughout the extension study. Study treatment will end when the patient dies, is lost to follow-up, withdraws informed consent, experiences sustained side-effects, has disease progression, or the sponsor discontinues the extension study. After the end of study visit is completed for the extension study, participants will be followed every 12 weeks for survival for up to 3 years following entry into the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma (cancer that begins in cells that line certain internal organs and that have secretory properties) of the prostate, but not with neuroendocrine differentiation or of small cell histology
* Before chemotherapy for prostate cancer with regimen(s) containing paclitaxel or docetaxel
* Documented prostate-specific antigen (PSA) progression according to PSA working group eligibility criteria with a PSA greater than 5 nanogram per milliliter (ng/mL)
* Ongoing androgen deprivation with serum testosterone level of less than 50 nanogram per deciliter (ng/dL)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 2 (Karnofsky Performance Status greater than or equal 50 percentage)

Exclusion Criteria:

* Active or uncontrolled autoimmune disease that may require corticosteroid therapy
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension
* Clinically significant heart disease as evidenced by a myocardial infarction in the past 12 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease (participants with a history of atherosclerotic vascular disease requiring coronary or peripheral artery bypass surgery may be enrolled provided the surgery occurred at least 2 years before to enrollment and after consultation with a cardiologist to insure that the disease is stable)
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (3):
- United States (2):
  - San Francisco, California
  - New York, New York
- Sutton, United Kingdom

REFERENCES:
- [Derived] Danila DC, Anand A, Sung CC, Heller G, Leversha MA, Cao L, Lilja H, Molina A, Sawyers CL, Fleisher M, Scher HI. TMPRSS2-ERG status in circulating tumor cells as a predictive biomarker of sensitivity in castration-resistant prostate cancer patients treated with abiraterone acetate. Eur Urol. 2011 Nov;60(5):897-904. doi: 10.1016/j.eururo.2011.07.011. Epub 2011 Jul 14. PMID 21802835
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov/
- See also: PROSTATE CANCER — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 5 participants in the Extension Study received treatment until they experienced progressive disease.
Groups:
- Abiraterone Acetate (Main Study): Abiraterone acetate 1000 milligram (mg) capsule or tablet was administered orally, once daily continuously in 28-day cycles up to 12 cycles, along with prednisone/prednisolone 5 mg tablet orally twice daily or dexamethasone 0.5 mg tablet orally once daily.
- Arbitarone Acetate (Extension): Participants who received abiraterone acetate 1000 milligram (mg) capsule or tablet orally, once daily continuously in 28-day cycles up to 12 cycles, along with prednisone/prednisolone 5 mg tablet orally twice daily or dexamethasone 0.5 mg tablet orally once daily in Main study, continued the same treatment until disease progression, death, or end of study (Week 148).
Period: Main Study
Arm/Group | Abiraterone Acetate (Main Study) | Arbitarone Acetate (Extension)
Started | 47 | 0
Completed | 11 | 0
Not Completed | 36 | 0
Not completed — Adverse Event | 11 | 0
Not completed — Symptomatic Deterioration | 1 | 0
Not completed — Progressive Disease | 23 | 0
Not completed — Other | 1 | 0
Period: Between Main Study and Extension
Arm/Group | Abiraterone Acetate (Main Study) | Arbitarone Acetate (Extension)
Started | 11 | 0
Completed | 5 | 0
Not Completed | 6 | 0
Not completed — Did Not Enter Extension Phase | 6 | 0
Period: Extension
Arm/Group | Abiraterone Acetate (Main Study) | Arbitarone Acetate (Extension)
Started | 0 | 5
Completed | 0 | 0
Not Completed | 0 | 5
Not completed — Progressive Disease | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Abiraterone Acetate: Abiraterone acetate 1000 milligram (mg) capsule or tablet was administered orally, once daily continuously in 28-day cycle up to disease progression, death, or end of study (Week 148), along with prednisone/prednisolone 5 mg tablet orally twice daily or dexamethasone 0.5 mg tablet orally once daily.
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Prostate Specific Antigen (PSA) Response at Week 12
Description: The PSA response was evaluated according to Prostate-Specific Antigen Working Group (PSAWG) criteria, which was, greater than or equal to 50 percent decrease in PSA from Baseline and confirmed by subsequent measurement at least 4 weeks later.
Time Frame: Baseline, Week 12
Population: The Intent-to-treat (ITT) population included all the participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
percentage of participants | 36.2 [22.7 to 51.5]

2. Secondary Outcome: Percentage of Participants With Confirmed Prostate Specific Antigen (PSA) Response
Description: as for outcome 1
Time Frame: Baseline up to Week 12
Population: The Intent-to-treat (ITT) population included all the participants who were enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
percentage of participants | 44.7 [30.2 to 59.9]

3. Secondary Outcome: Percentage of Participants With Confirmed Objective Tumor Response as Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: The objective tumor response was defined as the percentage of participants achieving a complete (CR) or partial response (PR) on tumor response assessed as per RECIST. The CR was disappearance of all lesions. The PR was at least a 30 percent decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the Baseline sum LD.
Time Frame: Baseline until first documented disease progression or end of study visit (Week 148; assessed on Day 1 of Cycle 4, 7, 10, and thereafter Day 1 of each cycle)
Population: The ITT population included all the participants who were enrolled into the study. Here 'N' (number of participants analyzed) signifies evaluable participants with measurable disease (the presence of at least one measurable lesion) at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 23
percentage of participants | 26.1 [10.2 to 48.4]

4. Secondary Outcome: Time to PSA Progression
Description: The time to PSA progression was the interval from the date of the first dose of abiraterone acetate to the date of PSA progression as defined by the PSAWG criteria. PSA progression was defined as a 50 percent increase over the nadir PSA value, increase in the PSA level by at least 5 nanogram per milliliter (ng/mL), and confirmed by second consecutive measurement.
Time Frame: Baseline until first documented disease progression or up to end of study (Week 148; assessed on Days 1, 8 of Cycle 1, thereafter Day 1 of each Cycle)
Population: The ITT population included all the participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
days | 169 [113 to 281]

5. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response was the time between the date of first PSA response (greater than or equal to 50 percent decline from Baseline) and the date of PSA progression as defined by the PSAWG. PSA progression was defined as a 50 percent increase over the nadir PSA value, increase in the PSA level by at least 5 nanogram per milliliter (ng/mL), and confirmed by second consecutive measurement.
Time Frame: as for outcome 4
Population: The ITT population included all the participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
days | 169 [141 to 262]

6. Secondary Outcome: Progression Free Survival Time
Description: Progression Free Survival was defined as the interval from the date of the first dose of abiraterone acetate to the date of death or date of progressive disease (PD) as assessed by RECIST criteria. PD was at least 20 percent increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline until first documented disease progression or death or up to end of study (Week 148; assessed on Day 1 of each cycle)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 23
days | 457 [163 to 712]

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from the date of the first dose of abiraterone acetate to the date of death.
Time Frame: Baseline until death, or end of study (Week 148)
Population: The ITT population included all the participants who were enrolled into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
days | 380 [311 to 457]

8. Secondary Outcome: Shift From Baseline in Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score at Post-dose (Week 148)
Description: The ECOG performance status score ranges from 0 to 5 where 0=fully active, perform all pre-disease activities without restriction; 1=restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature; 2=ambulatory, capable of self-care, unable to carry out any work activities, up and about more than (>) 50 percentage of waking hours; 3=capable of limited self-care, confined to bed or chair >50 percentage of waking hours; 4=completely disabled, not capable of any self-care, totally confined to bed or chair; and 5=dead.
Time Frame: Baseline until first documented disease progression or up to end of study (Week 148; assessed on Day 1 of each cycle)
Population: The ITT population included all the participants who were enrolled into the study.
Measure: Number; unit: participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 47
participants
  Baseline, ECOG 0 | 16
  Baseline, ECOG 1 | 27
  Baseline, ECOG 2 | 4
  Best Post-Baseline. ECOG 0 | 25
  Best Post-Baseline. ECOG 1 | 19
  Best Post-Baseline. ECOG 2 | 3

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 30 days after the last dose of study medication
Arm/Group | Abiraterone Acetate
Serious Adverse Events (participants affected / at risk) | 27/47
Other Adverse Events (participants affected / at risk) | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=47)
Anaemia (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Pitting oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1
Transaminases increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=47)
Anaemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 25
Oedema peripheral (General disorders) | 13
Cellulitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 8
Contusion (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood albumin decreased (Investigations) | 4
Blood creatine increased (Investigations) | 3
Blood sodium increased (Investigations) | 3
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 6
White blood cell count decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 13
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Groin pain (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 4
Haematuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less